CLINICAL TRIAL: NCT04853771
Title: The Effect of Progressive Muscle Relaxation Exercise Training Given to Pregnant Women With Restless Leg Syndrome on Symptom Severity, Sleep and Quality of Life
Brief Title: The Effect of Progressive Muscle Relaxation Exercise Training Given to Pregnant Women With Restless Leg Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Pinar Akbas, Expert Nurse, Doctoral student, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAkbas
Record Dates: First submitted 2021-04-04; First posted 2021-04-21 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Restless Legs Syndrome
Keywords: restless legs sendrome; progressive muscle relaxation exercise; quality of life; sleep hygiene
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: Research, single -centered , stratified randomization (hafif-moderate, severe-very severe ) with a pre-test and post-test control group parallel randomized control with experimental was designed as an operation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment (Experimental): 28-29. Between the weeks of gestation, one-time progressive muscle relaxation exercise training prepared by the researcher will be given to the pregnant women. Exercise will be demonstrated in training. Later, pregnant women will be asked to explain and practice the exercise. Women will be repeated until they do the exercise completely correctly (Check-list 1). After the training, pregnant women will be asked to do progressive relaxation exercises at least 3 times a week (every other day). With the progressive muscle relaxation exercise daily follow-up schedule prepared by the researcher, the pregnant women will be followed for 8 weeks and weekly reminders will be made (via whatsapp® or text message). The final test application (36-37 weeks) will be done online at the end of 8 weeks to the pregnant women. In pre-test and post-test applications, RLS Severity Rating Scale form, Johns Hopkins Restless Leg Syndrome Quality of Life Scale and Pittsburg Sleep Quality Index will be used.
  Interventions: Behavioral: progressive muscle relaxation exercise training
- control (No Intervention): No intervention will be applied to pregnant women, other than the routine training given in the pregnancy school. In the maternity school, training is given on physiological and psychological changes that occur during pregnancy, baby care, postpartum period, family planning. However, pregnant women are not given any information about RLS, coping methods, creating a healthy lifestyle, and progressive muscle relaxation exercises. Final test application to pregnant women; 36-37. It will be held online between weeks. In pre-test and post-test applications, RLS Severity Rating Scale form, Johns Hopkins Restless Leg Syndrome Quality of Life Scale and Pittsburg Sleep Quality Index will be used.

INTERVENTIONS:
Behavioral: progressive muscle relaxation exercise training — Progressive muscle relaxation exercises (PKGE); 16 large muscles (right hand and forearm, right upper arm, left hand and forearm of left arm, left upper arm, forehead, upper cheek and nose, chin, neck, abdomen, upper right arm, which people can do on their own after learning) leg, right calf, right foot, left upper leg, left thigh and left foot), followed by the contraction and then relaxation and accompanied by deep breathing, is a preferred method for reducing pain, anxiety and depression in individuals.The relaxation will be required to take 10-20 before stretching the next muscle group. In this way, the muscle groups in the hands, arms, neck, shoulder, chest, abdomen, hips, feet and fingers, face and the whole body will be voluntarily stretched and relaxed, and pregnant women will be relieved.
  Arms: experiment

SUMMARY:
Restless Leg Syndrome (RLS) is a sensory-motor problem characterized by an uncomfortable and unpleasant feeling that causes a strong and overwhelming desire to move the legs, usually during periods of inactivity during sleep.It is reported that pregnancy is an important risk factor in the onset and worsening of RLS.Individuals with RLS avoid social activities, often experience psychiatric problems such as depression, anxiety disorders, and chronic sleep disorders. Therefore, restless leg syndrome significantly affects daily life and coping with these problems. Individuals with RLS initially undertake a variety of non-pharmacological practices to relieve symptoms.Progressive muscle relaxation exercises, reducing the level of epinephrine and norepinephrine in the blood and heart rate, reducing oxygen consumption, regulating metabolic rate, lowering blood pressure, reducing muscle tension, preventing fatigue and restlessness, decreasing pain by increasing endorphin levels, increasing coping with pain and stress, It has many benefits such as improving sleep and quality of life.This study will be conducted to evaluate the effect of progressive muscle relaxation exercise training and follow-up given to pregnant women with restless leg syndrome on the severity of restless leg syndrome, quality of life associated with restless legs syndrome, and sleep quality.

DETAILED DESCRIPTION:
Restless Leg Syndrome (RLS) is a sensory-motor problem characterized by an uncomfortable and unpleasant feeling that causes a strong and irresistible desire to move in the legs, usually during periods of inactivity during sleep. Depending on cultural, environmental and genetic differences, the prevalence of RLS is reported to be the highest in North America and Europe, ranging from 5.5% to 11.6%, and this prevalence is reported to be between 1.0 and 7.5% in Asia. Turkey made society based on two studies in RLS prevalence of respectively 3.19% and 7% were found.

HBS 's with age, e increases from and in women has been reported from two times higher than that seen in man. The reason for its higher incidence in women has not been clearly explained, but it has been thought to be related to hormonal changes during pregnancy, menstruation and menopause. In a systematic review and meta-analysis study, it was reported that the prevalence of RLS in pregnant women worldwide is 21% and the symptoms are more common in the third trimester. In our country, g is reported to vary between midwives in HBS 19-26% incidence. In the study conducted by Neyal et al. (2015) in our country, it was found that 15.6% in the first trimester of pregnancy; 32.8 % in the second trimester ; It is reported that RLS symptoms are observed with a rate of 38.8% in the third trimester and the symptoms continue at a rate of 34.8% after birth. In the study conducted by Akbaş and Yaman Sözbir (2019), approximately half of the pregnant women (46.4%) had RLS symptoms and the RLS severity mean score of pregnant women with RLS was found to be 20.82 ± 6.61 . In the same study, the HBS of 49.1% of women with severe and very Siddiqui has been determined that there is live meat that fell to the severity of RLS increases quality of life reported and un.

Pregnancy is reported to be an important risk factor in the onset and worsening of RLS. It has been proven that the dopaminergic system plays an important role in the pathogenesis of RLS . Iron acts as a cofactor in the synthesis and formation of dopamine and normal dopamine production is impaired in iron deficiency. It is reported that increased iron need and anemia during pregnancy triggers RLS and the problem gets worse in the third trimester of pregnancy. In addition, vitamin D and folate increase dopamine synthesis and are reported to be protective of dopaminargic neurons and the brain against metabolite toxins. Studies have shown that iron , folate, and vitamin D deficiency cause restless leg syndrome. In addition, increasing estrogen, progesterone and prolactin levels during pregnancy accelerate the appearance of symptoms, especially in the third trimester. It has been reported that estrogen inhibits the synthesis and release of dopamine during pregnancy and progesterone increases neuronal excitability, leading to frequent hyper- reflexes and periodic leg movements and RLS during pregnancy. After birth, with the rapid increase of prolactin hormone, symptoms begin to improve.

Individuals with RLS avoid social activities, often experience psychiatric problems such as depression, anxiety disorders, and chronic sleep disorders. Therefore, restless leg syndrome significantly affects daily life and coping with these problems . HBS to relieve symptoms of various individuals who initially non-pharmacological located in the application s . However, it may be necessary to benefit from pharmacological treatment in cases with severe RLS. However, the use of drugs in pregnant women may be inconvenient. A standard drug therapy has not been determined for the treatment of RLS in pregnant women and the number of drugs that can be used is limited. Because most drugs have been used according to the evidence of non-pregnant patients and controlled studies in the treatment of RLS during pregnancy are insufficient. Therefore, GeBa steel during treatment of RLS in terms of drug therapy with the benefits of fetal compromise between the advantages/disadvantages of evaluation and decision making in this regard is necessary . However, during the treatment of RLS in pregnancy, the effect of drugs on the fetus , especially putting njenital me lformasyo considering the possibility should be taken.

The purpose of progressive relaxation exercises; It is to learn to feel the difference between tension and looseness in our body and to relax by ourselves in our daily life. For this purpose, the most widely used muscle groups, hands, arms, neck, shoulders, face, chest, abdomen, hips, feet and fingers were run . This method, which is applied in the form of stretching and relaxing the muscles , enables people to learn where their muscles are, what they have become during tension, and the difference when this tension disappears.

Progressive muscle relaxation exercises, reducing the level of epinephrine and norepinephrine in the blood and heart rate, reducing oxygen consumption, regulating metabolic rate, lowering blood pressure, reducing muscle tension, preventing fatigue and restlessness, reducing pain by increasing endorphin levels, increasing coping with pain and stress, It has many benefits such as increasing the quality of sleep and life.

RLS, which increases in frequency during pregnancy, disrupts sleep quality and affects the quality of life as it increases fatigue in pregnant women. During the follow-up, care and counseling process performed by nurses during pregnancy, pregnant women should be evaluated for sleep disturbance, fatigue, anxiety and stress that may be caused by RLS and attempts should be made to increase the quality of life by solving problems in cases . At this point, it is especially important to teach how to deal with RLS or how to relieve symptoms . In this context, progressive muscle relaxation exercises, which have many benefits and can be applied by nurses, should be taught to pregnant women during the routine follow-up and care process, and the use of relaxation exercises should be provided both at home and in clinics.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 20-34
* 25-28 days of her pregnancy. being in weeks of gestation
* Not having any chronic disease
* Not having any psychiatric illness
* Not being pregnant at risk
* Not having any communication problems (mental, auditory, visual, etc.)

Exclusion Criteria:

* Pregnancy does not do the post-test applications
* Failure to do progressive muscle relaxation exercises 2 times in a row
* Willing to leave research
* Other complications during pregnancy
* Hospitalization of the woman
* Early termination of pregnancy
* Not reaching pregnant woman during follow-up

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Restless Legs Syndrome Severity | Change from Baseline RLS Severity at 8 weeks
  Measurements will be made using the RLS Severity Rating Scale.
quality of life associated with restless legs syndrome | Change from Baseline Quality of Life at 8 weeks
  Measurements will be made using the Johns Hopkins Restless Leg Syndrome Quality of Life Scale.
quality of sleep associated with restless legs syndrome | Change from Baseline Quality of Sleep at 8 weeks
  Measurements will be made using the Pittsburg Sleep Quality Index.

CONTACTS AND LOCATIONS:
Overall Officials: Şengül YAMAN SÖZBİR, PhD, Principal Investigator — Gazi Universty
Locations (1):
- Karabük Training and Research Hospital, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Akbas P, Yaman Sozbir S. The effect of progressive muscle relaxation exercise on the intensity of symptoms and quality of sleep and quality of life in pregnant women with restless leg syndrome. Patient Educ Couns. 2023 Aug;113:107768. doi: 10.1016/j.pec.2023.107768. Epub 2023 Apr 28. PMID 37146530